CLINICAL TRIAL: NCT02223689
Title: Evaluation of SkinAffix as a Topical Emergency Room Department Skin Incision Adhesive
Brief Title: Evaluation of Skin Affix in the Emergency Room
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R14-008
Record Dates: First submitted 2014-03-27; First posted 2014-08-22 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2016-02

CONDITIONS: Wounds
Keywords: SkinAffix
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skin Affix (Experimental): Surgical adhesive
  Interventions: Procedure: Skin Affix

INTERVENTIONS:
Procedure: Skin Affix

SUMMARY:
Effectiveness of a surgical adhesive on wounds found in Emergency Medicine.

DETAILED DESCRIPTION:
Subjects were approached for recruitment in the ED when discussing closure options by the physician. Only subjects deemed appropriate for skin glue closures by their treating physician were approached.Subjects were followed at 48 hours post-procedure, 5-10 days, and at 14 days following the ED visit.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 5 years of age
* Requires the use of a surgical skin adhesive
* Informed consent signed

Exclusion Criteria:

* Sensitivity to topical adhesive products or formaldehyde
* Hx keloid formation, hypotension, diabetes, blood clotting disorders
* Wound infections
* mucosal surfaces or skin exposed to body fluids

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Schrock, MD, Principal Investigator — Metro Hospital
Locations (1):
- MetroHealth System, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Skin Affix: Surgical adhesive (Skin Affix) applied during wound closure in ED
Period: Overall Study
Arm/Group | Skin Affix
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Skin Affix: Surgical adhesive
  Skin Affix
Arm/Group | Skin Affix
Number analyzed (Participants) | 35
Age, Continuous [Mean (Full Range); unit: years] | 33.1 [7 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 24
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Wound Closure at Discharge
Description: Wounds remained closed following application of Skin Affix
Time Frame: 14 days
Measure: Number; unit: percent of participants
Arm/Group | Skin Affix
Number analyzed (Participants) | 35
percent of participants | 100

2. Secondary Outcome: Change in Pain Following Application
Description: Any 1 point decrease, increase, or no change in pain was measured on a scale--0 =no pain = 5 most pain.
Time Frame: 15 minutes Post Application
Population: Participants were asked 15 min after application to rate any change in pain as decreased, increased or no change.
Measure: Number; unit: percent of participants
Groups:
- Change in Pain Following Application: Pain assessed through a pain score 0-5. 0 = no pain, 5 = highest pain.
Arm/Group | Change in Pain Following Application
Number analyzed (Participants) | 35
percent of participants
  Increase in Pain | 8.6
  Decrease in Pain | 22.9
  No change in Pain | 57.1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Skin Affix
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 9/35
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Skin Affix (N=35)
Procedural bleeding (Surgical and medical procedures) | 3 (3)
Dihiscence (Surgical and medical procedures) | 4 (4)
Infection (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No